CLINICAL TRIAL: NCT02691897
Title: The Effects of Melatonin on Serum Glucose Levels of Patients With Type 2 Diabetes Mellitus
Brief Title: Melatonin's Effects on Treatment Of Diabetes Mellitus
Acronym: METOD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal Medicine & Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-93-7817
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Melatonin; Blood Glucose; Therapeutics; Pineal gland
MeSH Terms: conditions — Diabetes Mellitus | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Melatonin 3mg once daily at bedtime
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo 1 tablet once daily at bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin 3mg once daily at bedtime
  Arms: Melatonin
Drug: Placebo — Placebo 1 tablet once daily at bedtime
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the efficacy and safety of melatonin in control of blood sugar in patients with type 2 diabetes mellitus (DM).

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a major public health problem with increasing worldwide incidence. The main causes for increase in incidence of DM are inactivity, obesity and changes of dietary habits. Investigators think that the changes in the awake-sleep cycle may also contribute to higher incidence of DM in recent years. Melatonin is an important component of the circadian system. Numerous experimental studies have demonstrated that melatonin has many beneficial actions.Melatonin is a potent antioxidant, reduces inflammatory process, lowers blood pressure, improve lipid profiles. Collectively, these data suggest that melatonin may be useful in control of blood sugar in patients with DM.

The aim of this study is to assess the efficacy of melatonin in control of blood sugar in patients with type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus diagnosed by an endocrinologist for more than six months
* FBS=120-160mg/dl
* HbA1C<8%

Exclusion Criteria:

* Melatonin sensitivity
* Impaired fasting glucose (IFG)
* Impaired glucose tolerance (IGT)
* Under Insulin therapy
* Pregnancy
* Lactation
* Diabetic autonomic neuropathy and orthostatic hypotension
* Renal failure (Creatinin>1.5mg/dl)
* Diabetic retinopathy
* Diabetic nephropathy
* Malignancy
* Alcohol use
* Liver disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Fasting blood sugar (FBS) | 3 months
HbA1c | 3 months

SECONDARY OUTCOMES:
Serum Insulin | 3 months
Weight (Body mass index) | 3 months
Waist circumference | 3 months
Serum aminotransferases | 3 months
Number of patients with adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Bagheri Lankarani, M.D., Study Chair — Health Policy Research Center, Shiraz University of Medical Sciences; Mesbah Shams, M.D., Principal Investigator — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Payam Peymani, Principal Investigator — Health Policy Research Center, Shiraz University of Medical Sciences
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No